# Goodwill of Central Texas: Fatherhood Works Healthy Marriage and Responsible Fatherhood Program Evaluation

**Study Protocol** 

**January 9, 2025** 

Clinicaltrials.gov ID: NCT05292963

#### PROGRAM BACKGROUND

#### 1. PROGRAM SUMMARY

Please provide a brief summary of your grant project including the needs to be addressed, the services provided, and the population served.

Children's healthy physical, emotional, and social development is strongly influenced by their family circumstances. Research has shown that engaged, supportive fathers and father figures can promote children's healthy development, while poverty can have significant long-term negative impacts on child development and educational attainment. Fathers and families in the Central Texas area, which includes Travis, Williamson, Hays, and Bastrop counties, face an increasingly high cost of living and rising poverty rates that make it difficult to meet their basic needs. The Central Texas area has a need for services that support low-income fathers to achieve greater economic stability, strengthen relationships, and be effective, nurturing parents.

Goodwill of Central Texas (GCT) aims to help low-income (<200% FPL) fathers and father figures 18 years of age or older in the Austin metropolitan area fulfill their roles and responsibilities through the Fatherhood Works Program (FWP). All FWP participants will receive a range of support services tailored to individuals' needs related to financial planning, career counseling, job search assistance, and occupational skills training. For delivering primary curriculum, GCT will partner with Any Baby Can, an experienced local nonprofit parenting skills training provider, to offer the evidence-based, skills-based *Nurturing Fathers* (*NF*) curriculum with workshops designed to teach parenting and nurturing skills to men. GCT will offer the *NF* curriculum in both virtual and in-person formats. GCT will also partner with SAFE Alliance, another local nonprofit training provider, to virtually offer the *Creating a Safe Home* primary curriculum designed to promote safe home environments.

#### 2. EVALUATION GOALS

Please briefly describe key goals of your evaluation and what you hope to learn below.

The key goal of this descriptive evaluation is to assess the extent to which participation in the Fatherhood Works Program is positively associated with improved attitudes and behaviors among low-income fathers and father figures in Central Texas. Research questions will focus on whether attitudes and behaviors related to parenting, partner relationships, and employment change after participation in primary program services.

#### 3. EVALUATION ENROLLMENT

Please provide the expected start and end dates for program and evaluation enrollment using the tables below.

| IMPLEMENTATION EVALUATION Please leave blank if not conducting an implementation study. | | |
|---|---|---|
| | Program Enrollment Study Enrollment | |
| Start Date | 05/01/2021 | 05/01/2021 |
| End Date | 07/15/2025 | 07/15/2025 |

## **Definition**

Program implementation metrics using data from nFORM (e.g., workshop hours received, enrollment, retention, etc.), site visit findings, CQI process findings

Same as program enrollment

| Please leave blank if not conducting a descriptive outcome evaluation. | | |
|---|---|---|
| | Program Enrollment Study Enrollment | |
| Start Date | 05/01/2021 | 05/01/2021 |

**DESCRIPTIVE EVALUATION** 

End Date 07/15/2025 06/15/2024

Definition Eligible low-income fathers and father figures in the Central Texas area, 18 All participants who cons

figures in the Central Texas area, 18
years of age or older, with children
under the age of 24

All participants who consent to be part
of the evaluation study

## 4. EVALUATION TIMELINE

Please include a timeline for key activities of the evaluation below.

| Evaluation Activity | Start Date | End Date |
|---|---|---|
| Additional evaluation staff hiring and onboarding | 1/15/2021 | 2/15/2021 |
| Evaluation staff training | 1/22/2021 | 2/20/2021 |
| Evaluation kickoff meeting and orientation with all program staff | 2/10/2021 | 2/10/2021 |
| IRB training and certification by all program and evaluation staff | 10/1/2020 | 3/09/2021 |
| Development and submission of descriptive evaluation plan document | 7/25/2022 | 8/25/2022 |
| Evaluation Tools Development | 10/1/2020 | 10/15/2021 |
| IRB Approval | 3/22/2021 | 3/29/2021 – initial<br>approval |

| | | 4/6/2022 – amendment approval |
|---|---|---|
| CQI Team Formed and Meeting bi-weekly | 5/20/2021 | 7/1/2025 |
| Training for CQI Team | 3/15/2021 | 3/28/2021<br>Ongoing as needed |
| Training for all Program Staff on Research Methods and process | 3/15/2021 | 4/12/2021<br>Ongoing as needed |
| Implementation Evaluation Data Collection | 4/15/2021 | 6/15/2025 |
| Evaluation Program Staff Training | 3/15/2021 | Ongoing as needed |
| Preliminary Implementation Report Submitted | 6/31/2022 | 6/31/2022 |
| Descriptive Study Data Collection | | |
| - Randomization | - | - |
| - Baseline | 4/15/2021 | 3/31/2024 |
| - Post Test | 7/8/2021 | 5/31/2024 |
| - Follow-up | 4/15/2022 | 6/15/2025 |
| Final Implementation Report Submitted | 9/1/2025 | 9/29/2025 |
| Final Report Submitted | 9/1/2025 | 9/29/2025 |

Commented [JL1]: Is this date correct?

# **EVALUATION PLAN**

# 1. RESEARCH QUESTIONS

## 1.1. OVERVIEW OF RESEARCH QUESTIONS

Research questions in this study are framed by a descriptive evaluation design that will be used to measures changes in participant outcomes after participation in the Fatherhood Works Program. Analyses will measure the differences in primary and secondary outcomes from orientation to one year after program enrollment. Primary outcomes refer here to changes in parenting and co-parenting *behaviors*. Secondary outcomes refer here to the *attitudes* that theoretically facilitate and reflect behaviors. Implementation analyses seek to demonstrate whether or not participants are receiving the intended amounts of FWP services.

| No | Research Question | Implementation or Outcome? |
|---|---|---|
| 11 | To what extent is the <i>Nurturing Fathers</i> curriculum offered to and received by program participants? | Implementation |
| 12 | To what extent are additional primary workshops offered to and received by program participants? | Implementation |
| 13 | To what extent did the CQI team carry out the steps in the CQI plan each program year? | Implementation |
| R1 | How did <b>parenting behavior</b> measures change from program enrollment to 1 year after enrollment? | Primary Outcome |
| R2 | How did <b>parenting attitude</b> measures change from program enrollment to immediately following program completion? | Secondary Outcome |
| R3 | How did <b>co-parenting behavior</b> measures change from program enrollment to 1 year after enrollment? | Primary Outcome |
| R4 | How did <b>employment attitude</b> measures change from program enrollment to 1 year after enrollment? | Secondary Outcome |

## 1.2. OUTCOME RESEARCH QUESTIONS

For each <u>outcome research question</u> listed above, whether a descriptive or impact design, summarize the inputs (e.g., program components, program supports, implementation features, etc.), target population (e.g., the population for which the effect will be estimated) and the outcomes (e.g., child well-being, father-child engagement, etc.) that will be examined to answer the research question(s). Comparisons for descriptive evaluations may reflect circumstances before the grant, pre-treatment, or pre-determined benchmark from other studies with similar interventions.

| Question Number correspond to the number te | ntervention Program component or set of activities hat the evaluation will est or examine | Target Populatio n Population for which the effect of the treatment will be estimated | Comparison What the intervention will be compared to (e.g., pre- intervention for descriptive designs) | Outcome Changes that are expected to occur as a result of the intervention | Confirmatory or Exploratory? Confirmatory: those upon which conclusions will be drawn Exploratory: those that may provide additional |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

| | | | | | suggestive<br>evidence |
|---|---|---|---|---|---|
| R1 | Primary program services which include: Nurturing Fathers parenting course, Creating a Safe Home domestic violence seminar, and a Workforce Advancement workshop | Low-<br>income<br>fathers/<br>father<br>figures<br>who are<br>18+ years<br>of age with<br>children up<br>to 24<br>years | Pre-<br>intervention<br>outcome<br>scores | Participants will report improved parenting behaviors 1 year after enrolling in FWP primary services | Confirmatory |
| R2 | Primary program services which include: Nurturing Fathers parenting course, Creating a Safe Home domestic violence seminar, and a Workforce Advancement workshop | Low-<br>income<br>fathers/<br>father<br>figures<br>who are<br>18+ years<br>of age with<br>children up<br>to 24<br>years | Pre-<br>intervention<br>outcome<br>scores | Participants will report improved parenting attitudes immediately following FWP primary services | Confirmatory |
| R3 | Primary program services which include: Nurturing Fathers parenting course, Creating a Safe Home domestic violence seminar, and a | Low-income fathers/ father figures who are 18+ years of age with children up to 24 years | Pre-<br>intervention<br>outcome<br>scores | Participants will report improved co- parenting behaviors 1 year after enrolling in FWP primary services | Confirmatory |

| | Workforce<br>Advancement<br>workshop | | | | |
|---|---|---|---|---|---|
| R4 | Primary program services which include: Nurturing Fathers parenting course, Creating a Safe Home domestic violence seminar, and a Workforce Advancement workshop | Low-income fathers/ father figures who are 18+ years of age with children up to 24 years | Pre-<br>intervention<br>outcome<br>scores | Participants will report improved employment attitudes 1 year after enrolling in FWP primary services | Confirmatory |

## 2. BACKGROUND

For each <u>outcome research question listed in 1.1</u>, whether descriptive or impact design, briefly summarize the previous literature or existing research that informs the stated research question and how the evaluation will expand the evidence base. Explain why the research questions are of specific interest to the program and/or community. Only a short summary paragraph description is needed below. Additional documentation, such as a literature review, may be appended to this document.

| Research<br>Question<br>Topic | Existing Research | Contribution to the Evidence Base | Interest to the<br>Program and/or<br>Community |
|---|---|---|---|
| R1 | Nurturing Fathers is an evidence-based curriculum that has been proven effective at building skills needed for healthy family relationships and child development. | Determine to what extent participation in a program that uses Nurturing Fathers curriculum, in combination with other workshop programming, is associated with changes in parenting behaviors among lowincome fathers and father figures in Central Texas. | Healthy parenting<br>behaviors support<br>children to achieve more<br>positive outcomes, both<br>short- and long-term,<br>and promote adult<br>wellbeing. |
| R2 | Nurturing Fathers is an evidence-based curriculum that has | Determine to what extent participation in a program that uses Nurturing | Healthy parenting attitudes facilitate healthy parenting |

| | been proven effective at<br>building skills needed<br>for healthy family<br>relationships and child<br>development. | Fathers curriculum, in combination with other workshop programming, is associated with changes in parenting attitudes among lowincome fathers and father figures in Central Texas. | behaviors, which in turn<br>support children to<br>achieve more positive<br>outcomes, both short-<br>and long-term, and<br>promote adult wellbeing. |
|---|---|---|---|
| R3 | Nurturing Fathers is an evidence-based curriculum that has been proven effective at building skills needed for healthy family relationships and child development. | Determine to what extent participation in a program that uses Nurturing Fathers curriculum, in combination with other workshop programming, is associated with changes in co-parenting behaviors among lowincome fathers and father figures in Central Texas. | Healthy co-parenting<br>behaviors support<br>children to achieve more<br>positive outcomes, both<br>short- and long-term,<br>and promote adult<br>wellbeing. |
| R4 | Nurturing Fathers is an evidence-based curriculum that has been proven effective at building skills needed for healthy family relationships and child development. | Determine to what extent participation in a program that uses Nurturing Fathers curriculum, in combination with other workshop programming, is associated with changes in employment attitudes among lowincome fathers and father figures in Central Texas. | Healthy employment<br>attitudes support children<br>to achieve more positive<br>outcomes, both short-<br>and long-term, and<br>promote adult wellbeing. |

## 3. LOGIC MODEL

Clearly demonstrate how the research question(s) (and the related implementation features and/or participant outcomes) link to the proposed logic model and the theory of change for the program. You may append a copy of your logic model to this document.

The appended logic model specifies a theory of change for delivering virtual and in-person primary services and standard support services as part of the Fatherhood Works Program. Service delivery processes specified in the model are linked to the desired outcomes for healthy family relationships. Model specification incorporates a descriptive study design to measure change in primary and secondary participant outcomes from program enrollment to one year after enrollment.

<u>Service delivery processes</u>: Key aspects of service delivery processes in the theory of change—goals, inputs, activities, and outputs—articulate the experiences that are designed to solve specific problems for those who agree to participate in the Fatherhood Works Program. Solving each problem identifies three broad service delivery goals to maximize participation benefits for study groups as explained below:

- Goal 1 Deliver primary curricula workshops to Fatherhood Works Program participants: Project participants will be offered three primary curricula through Goodwill of Central Texas and their facilitation partner Any Baby Can, in combination with support services and case management. The Nurturing Fathers curriculum will help to develop participants' skills and healthy attitudes to engage in healthy parenting and co-parenting behaviors. The Creating a Safe Home seminar will help to build participant knowledge about domestic violence and child neglect to reduce these behaviors. The Workforce Advancement workshop will help to develop participants' job search skills and increase to the likelihood of securing stable, gainful employment. Participant engagement in the primary curricula and local evaluation surveys will take place after receiving the FWP orientation and providing project staff with informed consent to participate in study activities.
- Goal 2 Deliver support services to Fatherhood Works Program participants: Project
  participants will be offered support services, including case management, transportation
  supports, and referrals to additional services within and external to Goodwill. These support
  services are intended to increase the likelihood that participants will benefit from primary
  services and to reduce barriers to program retention.
- Goal 3 Conduct Continuous Quality Improvement (CQI) efforts to ensure full implementation of program services: Reports prepared and presented to the CQI Team by evaluators in the CQI process will use a series of performance indicators to track key outputs over time to identify any primary or support FWP services delivered to study groups that might fall short of the intended amounts to be offered (i.e., fidelity standards) and received (i.e., dosage thresholds) by them. The CQI Team will then work with project staff to develop and implement performance interventions to address any outputs that need improvement to ensure the services offered to, and received by, participants meet the intended amounts by the end of each program year.

<u>Desired Outcomes</u>: Outcomes specified in the logic model theorize the primary and secondary outcomes that are desired for program participants after they receive primary and support services. Secondary outcomes are the improved attitudes that facilitate and reflect participant engagement in healthy parenting and employment behaviors. Primary outcomes are the healthier parenting and co-parenting behaviors exhibited by participants that ultimately define the benefits of Fatherhood Works Program participation.

#### 4. HYPOTHESES

For each specified research question, state the hypothesized result(s) and briefly describe why these results are anticipated.

| Research Question | Hypothesized Result |
|---|---|
| R1 | Participants will report <b>healthier parenting behavior</b> one year after enrolling in the Fatherhood Works Program. |
| R2 | Participants will report <b>healthier parenting attitudes</b> immediately following the Fatherhood Works Program. |
| R3 | Participants will report <b>healthier co-parenting behavior</b> one year after enrolling in the Fatherhood Works Program. |
| R4 | Participants will report <b>healthier employment attitudes</b> one year after enrolling in the Fatherhood Works Program. |

# 5. RESEARCH DESIGN

For each research question, briefly describe why the research design proposed will answer each research question(s). State whether the proposed evaluation is a descriptive or impact evaluation and justify why the proposed research design is best suited to answer the research question(s).

| Research Question | Design | Justification |
|---|---|---|
| R1 | For this descriptive evaluation, healthy parenting behavior will be measured at the time of program enrollment and one year after program enrollment, and analyses will determine if changes in parenting behavior outcomes are statistically significant. | This study is interested in whether Fatherhood Works Program participation is associated with improved outcomes for participants, so a descriptive study is sufficient for measuring differences in participant outcomes over time. |
| R2 | For this descriptive evaluation, healthy parenting attitudes will be measured at the time of program enrollment and immediately following program completion, and analyses will determine if changes in parenting attitude outcomes are statistically significant. | This study is interested in whether Fatherhood Works Program participation is associated with improved outcomes for participants, so a descriptive study is sufficient for measuring differences in participant outcomes over time. |
| R3 | For this descriptive evaluation,<br>healthy co-parenting behavior will<br>be measured at the time of program<br>enrollment and one year after<br>program enrollment, and analyses | This study is interested in whether Fatherhood Works Program participation is associated with improved outcomes for participants, so a descriptive study is sufficient for |

| | will determine if changes in co-<br>parenting behavior outcomes are<br>statistically significant. | measuring differences in participant outcomes over time. |
|---|---|---|
| R4 | For this descriptive evaluation, healthy employment attitudes will be measured at the time of program enrollment and one year after program enrollment, and analyses will determine if changes in employment attitude outcomes are statistically significant. | This study is interested in whether Fatherhood Works Program participation is associated with improved outcomes for participants, so a descriptive study is sufficient for measuring differences in participant outcomes over time. |

#### 6. ONGOING GRANTEE AND LOCAL EVALUATOR COORDINATION

Describe how the grantee and local evaluator collaboratively worked together to identify the research question(s) and research design to ensure its feasibility and relevance. Describe how the grantee and local evaluator will continue to work together throughout the evaluation to proactively address unforeseen challenges as they arise and ensure the rigor and relevance of the evaluation and its findings. Describe how the grantee and local evaluator will coordinate dissemination efforts. Describe how these processes will occur while maintaining the independence of the evaluation.

The basis for ongoing coordination between GCT (the grantee) and MER (the local evaluator) is regular communication, by way of recurring meetings and daily interactions with embedded staff. Throughout the original proposal process, and now during the evaluation planning phase, MER worked with GCT to design a study with research questions that are appropriate to the intervention. MER guides the process, given our experience designing and running evaluations, and GCT provides expertise on their community, target population, and program/curricula specifics.

Recurring meetings will include a bi-weekly project CQI team meeting. Under the leadership of the Data Manager and Lead MER Evaluator, the CQI team reviews data from the nFORM and local evaluation systems to identify and mitigate implementation or data issues, and closely examine trends and accomplishments. This team includes GCT organizational and project leadership, the MER Evaluation team, and front-line staff representatives (e.g., Program Administrator, Career Case Managers).

In addition to CQI team meetings, overall project team meetings occur monthly (at a minimum), with project leaders across MER and GCT in attendance, to ensure the partnership remains strong and that coordination across organizations is on track. This recurring, ongoing meeting structure is conducive to close coordination, ensuring that challenges can be quickly addressed, and promising strategies can be efficiently maximized.

One of the key components of this coordination effort is the Data Manager, who is a MER employee, embedded with GCT. The Data Manager functions to bridge the gap between organizations. They will interact with GCT staff daily while completing their job duties and play a leadership role in the recurring meetings outlined above. See Section 8 below for more details about this role and others. Both the meetings and the roles outlined above will continue throughout

the entire project period, providing opportunities to ensure the rigor and relevance of the evaluation and its findings, and to discuss and coordinate dissemination efforts (which will also be shared across MER and GCT).

MER has experience operating prior evaluations using this exact process. Clearly outlining roles and responsibilities maintains the independence of the evaluation. That is, the evaluation team helps identify and illuminate areas of concern or improvement (for the program and the evaluation), but the program staff have responsibility for implementing improvements and providing direct services to participants. In this way, GCT and MER acknowledge our shared interest in and responsibility for a well-executed project and evaluation, but that MER is also an independent and external organization with a high level of integrity and is not responsible for, nor invested in, the specific outcomes of the program. This allows for close coordination without allowing for codependence, or for personal interests to influence evaluation findings.

#### 7. LEAD STAFF

Define the roles of lead staff for the evaluation from both organizations below.

| Name | Organization | Role in the Evaluation |
|---|---|---|
| Dr. Matthew Shepherd | Midwest Evaluation and Research | Principal Investigator |
| Charlene Brickner, MA | Midwest Evaluation and Research | Lead Evaluation Consultant and Evaluation Project Manager |
| Charlene Brickner, MA | Midwest Evaluation and Research | CQI Data Manager |

Articulate the experience, skills, and knowledge of the staff for the evaluation (including whether they have conducted similar studies in this field), as well as their ability to coordinate and support planning, implementation, and analysis related to a comprehensive evaluation plan.

Dr. Matthew Shepherd will serve as the Principal Investigator for this grant. As such, he has corporate responsibility for all evaluation activities. Dr. Shepherd has over 25 years' experience in program design and implementation, applied research, program evaluation, policy analysis, and evaluative technical assistance.

Charlene Brickner will serve as the Lead Evaluation Consultant and Evaluation Project Manager. She will lead the efforts to conduct a descriptive study <u>and</u> the Continuous Quality Improvement (CQI) process for the grant.

Charlene Brickner will also serve as the CQI Data Manager. Prior to joining MER, Ms. Brickner served as a research assistant with the Children's Learning Institute in Houston. The CQI Data Manager will work closely with the grantee and community partners on-site to complete data

collection and management activities for the impact study <u>and</u> a Continuous Quality Improvement (CQI) process.

#### 8. SAMPLE

#### 8.1. TARGET POPULATION(S)

For each target population identified in Section 1.2, please describe the target population(s), and explicitly state whether the population(s) differs from those who will be broadly served by the grant. Describe how the target population will be identified. Explicitly state the unit of analysis (e.g., non-residential father, unmarried couple).

| Description of<br>Target Population | How is the population different from those who will be broadly served by the grant? | How will the target population be identified? | Unit of<br>Analysis |
|---|---|---|---|
| Low-income fathers<br>and father figures<br>18 years of age or<br>older with children<br>24 years or<br>younger in the<br>Central Texas area | No difference, all<br>program participants<br>will be part of the<br>study sample | GCT and community partners will recruit potential participants in the target population. GCT will determine eligibility as part of their intake and screening process. | Father/Father<br>Figure |

## 8.2. METHODS TO PROMOTE SUFFICIENT PROGRAM PARTICIPATION

Please describe methods to promote sufficient program participation in the table below.

What methods will you use to ensure sufficient sample is recruited, enrolls, and participates in the program?

GCT and their community partners will recruit program participants, and GCT will provide incentives for workshop completion and successful program referrals. GCT has implemented organizational strategies to increase program enrollment, including prioritizing referrals to Fatherhood Works for all eligible walk-in clients. GCT also meets quarterly with its community partners to talk about progress toward meeting referral targets. The CQI process will address issues regarding program recruitment, enrollment, and completion to ensure targets are met.

| Who will be responsible for recruiting the evaluation sample? | The evaluation sample will not differ from the program population, in that all participants will be invited to participate in the evaluation. Enrollment into the evaluation will be conducted by the Data Manager who will conduct the informed consent process and proctor the baseline data collection efforts. |
|---|---|
| Please describe any incentives to be offered for program participation and/or completion and/or data collection and/or participation in the evaluation. | Program Participation – GCT will provide a series of incentives for workshop completion, employment retention, and successful referrals to the program, up to \$200. Evaluation Participation – The program participation incentive for reaching 100% of primary workshop hours includes exit survey completion. No incentive will be given for entrance survey completion. A \$50 Giftogram gift card will be given to participants who complete the 1-year follow- |

up survey.

## 9. DATA COLLECTION

## 9.1. CONSTRUCTS AND MEASURES

Clearly articulate the constructs of interest, measures to evaluate those constructs, and specific data collection instruments. Provide any information on the reliability and validity of the data collection instruments. For standardized instruments, you may provide the citation for the instrument.

| Construct | Measure | Instrument | Reliability and Validity |
|---|---|---|---|
| Parenting<br>Behavior | 1 item: hours spent with children in last 30 days (interval); 1 item: frequency reaching out to children (categories, 5-point scale); 7 items: frequency engaging in key behaviors (categories, 5-point scale) | nFORM Community-<br>Based Fathers Survey<br>(A2b, A2c, A5b: b-d, f-i) | nFORM |
| Parenting<br>Attitudes | 7 items: frequency of key attitudes (categories, 5-point scale) | nFORM Community-<br>Based Fathers Survey<br>(A3: a-g) | nFORM |

| Co-Parenting<br>Behavior | 11 items: frequency of agreement with key coparenting behaviors (interval, 5-point scale) | nFORM Community-<br>Based Fathers Survey<br>(A13: a-k) | nFORM |
|---|---|---|---|
| Employment<br>Attitudes | 2 items: level of agreement with attitudes related to acquiring a job and providing for a family. | OLLE (Online Local<br>Evaluation) Survey | Jurkiewicz, T. & Friedman, L. (2020). Impact Evaluation of The TYRO Champion Dads Project in Dallas, Texas: Final Impact Evaluation Report for Anthem Strong Families. Midwest Evaluation and Research. |

#### 9.2. CONSENT

Describe how and when program applicants will be informed of the study and will have the option of agreeing (i.e., consenting to) or declining to participate in the study.

Because the planned evaluation involves human subjects, GCT understands program implementation requires both IRB approval and participant informed consent. MER has an established relationship with Solutions IRB, having secured more than 20 IRB approvals and renewals for evaluations it has conducted during the past five years. IRB clearance will be submitted for approval and obtained during the planning period.

To secure informed consent, participants will attend an orientation / enrollment session (in person or virtual) where the Data Manager will describe the evaluation process and the risks and benefits of the project. An IRB-approved Q&A video can be played during orientation to provide more information about the evaluation study as needed. Those people that wish to participate in the evaluation will complete an informed consent process and sign an informed consent document / form. All participants will receive a copy of the consent form with contact information for evaluation staff and how to contact the IRB with any questions or to withdraw from the study. Informed consent will take place prior to the collection of evaluation data.

#### 9.3. METHODS OF DATA COLLECTION

If the evaluation will collect multiple waves of data, describe the timing of these waves below. When describing follow-up periods, specify whether the follow-up period will be post-baseline, post-random assignment, or post-program completion.

| Wave of Data Collection | Timing of Data Collection |
|-------------------------|---------------------------|

| (e.g., baseline, short-term follow-up, long-term follow-up) | |
|---|---|
| Baseline | Collected immediately following informed consent and study enrollment – during orientation session or first workshop |
| Post-test | Collected after the completion of the primary services programming – during the last workshop session or exit session – approximately 7 to 13 weeks after enrollment depending on delivery schedule |
| 1 year follow-up (post-baseline) | Collected approximately one year after study enrollment/baseline |

For each measure, describe how data will be collected detailing which data collection measures will be collected by which persons, and at what point in the programming or at what follow-up point.

| Survey | Timing of<br>Data<br>Collection<br>(baseline,<br>wave of data<br>collection) | Method of<br>Data<br>Collection | Who Is<br>Responsible<br>for Data<br>Collection? | Will Methods<br>or Collection<br>Procedures<br>Differ by<br>Study<br>Group? | Will data<br>access<br>require data<br>sharing<br>agreement? |
|---|---|---|---|---|---|
| On-Line<br>Local<br>Evaluation<br>(OLLE) and<br>nFORM<br>Baseline<br>Surveys | Baseline | Participant<br>self-enters<br>survey using<br>online data<br>collection<br>platform | Data Manager will proctor data collection and assist participants as necessary | No | N/A |
| OLLE and<br>nFORM Post-<br>Test Surveys | Post-Test<br>(approx. 7 to<br>13 weeks<br>after<br>enrollment) | Participant<br>self-enters<br>survey using<br>online data<br>collection<br>platform | Data Manager will proctor data collection and assist participants as necessary | No | N/A |

| OLLE 1 Year<br>Follow-up<br>Survey | 1 year after<br>enrollment /<br>baseline | Participant self-enters survey using online data collection platform and link – or – Phone interview data collection with evaluation staff | MER<br>Research<br>Staff/<br>participant<br>tracking team | No | N/A |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

#### 10. IRB/PROTECTION OF HUMAN SUBJECTS

Please describe the process for protection of human subjects, and IRB review and approval of the proposed program and evaluation plans. Name the specific IRB to which you expect to apply.

Solutions IRB, a private commercial Association for the Accreditation of Human Research Protection Programs Inc. (AAHRPP) fully accredited Institutional Review Board, will ensure that this study is approved before any research activities take place. MER has had 14 research studies approved by Solutions IRB over the past four years, has completed over 15 annual check-in reports, and has submitted timely amendments when changes to studies needed to take effect.

All submissions are completed online, so turnaround for a new study approval is between 24 to 72 hours, though the full approval process can take approximately one to two weeks depending on the number of questions and requested revisions that the IRB makes. In the IRB application submission, we will include descriptions of project staff, locations of study sites, the funding source, incentives, summary of activities, participant population, recruitment plans, risks and benefits, confidentiality of data, and the informed consent process along with all materials to be used in the study such as participant forms and surveys.

This project was submitted for IRB approval in early March 2021 and received official approval to begin enrollment and data collection in March 2021. Amendments to the original application were approved in April 2022 and will be submitted as necessary based on programmatic or evaluation changes.

#### 11.DATA

#### 11.1. DATABASES

For each database used to enter data, please describe the database into which data will be entered (i.e., nFORM and/or other databases), including both performance measure data you plan to use in your local evaluation and any additional local evaluation data. Describe the process for data entry (i.e., who will enter the data into the database).

| Database Name | Data Entered | Process for Data Entry |
|---|---|---|
| nFORM | Performance measurement data, local evaluation data | Entered directly by participants, and by program staff |
| Qualtrics | Local evaluation data, participant outcomes (OLLE survey) | Entered directly by participants, and by MER evaluation staff |

## 11.2. DATA REPORTING AND TRANSFER

For each database provided in the table above, please indicate the ability to export individual-level reports to an Excel or comma-delimited format and whether identifying information is available for linking to data from other sources.

| Database Name | Ability to Export Individual Reports? | What identifying information is available to facilitate linking to other data sources? |
|---|---|---|
| nFORM | Yes using Data Export function | nFORM ID, name, date of birth |
| Qualtrics | Yes, Excel or comma-<br>separated | nFORM ID, name, date of birth |

<sup>\*</sup> you may add rows by hitting the tab button, or right click and select insert row below

## 11.3. CURRENT SECURITY AND CONFIDENTIALITY STANDARDS

For each database provided in Section 11.1, please Indicate the ability to be able to encrypt data access during transit (for example, accessed through an HTTPS connection); be able to encrypt data at rest (that is, when not in transit), have in place a data backup and recovery plan; require all users to have logins and passwords to access the data they are authorized to view; and have current anti- virus software installed to detect and address malware, such as viruses and worms.

| Database Name | Ability to encrypt data during transit? | Ability to encrypt at rest? | Data<br>Backup and<br>Recovery<br>Plan? | Require all users to have logins and passwords? | Current Anti-<br>Virus Software<br>Installed? |
|---|---|---|---|---|---|
| Qualtrics | Yes | Yes | Yes | Yes | Yes |

Please describe any plans for study registration with an appropriate registry (e.g., clinicaltrials.gov, socialscienceregistry.org, osf.io, etc.).

MER will register this descriptive study with clinicaltrials.gov.